CLINICAL TRIAL: NCT00906334
Title: A Phase 2, Single-Arm Study To Assess The Efficacy and Safety Of 72-Hour Continuous Intravenous Dosing Of ON 01910.Na Administered Every Other Week in Myelodysplastic Syndrome Patients With Trisomy 8 or Classified as Intermediate-1, 2 or High Risk
Brief Title: Efficacy and Safety of ON 01910.Na in Myelodysplastic Syndrome (MDS) Patients With Trisomy 8 or Classified as Intermediate-1, -2 or High Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onconova 04-17; NCT01326377 (obsolete NCT alias)
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Trisomy 8; Intermediate-2 Risk Group; High-Risk Group; azacitidine; azacytidine; Vidaza; decitabine; Dacogen
MeSH Terms: conditions — Myelodysplastic Syndromes; Chromosome 8, trisomy | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 800 mg/m^2 ON 01910.Na (Experimental): 800 mg/m^2 ON 01910.Na administered as a continuous intravenous infusion (CIV) over 24 hours for 48 hours (i.e. 2 consecutive 24-hour infusions) every week for the first 3 weeks of 4-week cycle.
  Interventions: Drug: ON 01910.Na
- 1800 mg ON 01910.Na (Experimental): 1800 mg ON 01910.Na administered as a continuous intravenous infusion (CIV) over 24 hours for 72 hours (i.e., 3 consecutive 24-hour infusions) every 2 weeks for the first four 2-week cycles and every 4 weeks afterwards.
  Interventions: Drug: ON 01910.Na

INTERVENTIONS:
Drug: ON 01910.Na — The original dosing regimen was 800 mg/m^2 ON 01910.Na.
  Other Names: rigosertib
  Arms: 800 mg/m^2 ON 01910.Na
Drug: ON 01910.Na — Per Amendment 3 to the Protocol, the dosing regimen was changed to 1800 mg ON 01910.Na. Patients enrolled at the original dosing regimen could choose to remain in the original regimen or switch to the new regimen.
  Other Names: rigosertib
  Arms: 1800 mg ON 01910.Na

SUMMARY:
This study will explore the efficacy and safety of a regimen of ON 01910.Na as a 48-hour continuous intravenous infusion once a week for 3 weeks of a 4-week cycle in MDS patients with Trisomy 8 or classified as Intermediate-1, -2 or High Risk who are not responding to current therapeutic options. The rationale for this trial is based upon data from laboratory studies with ON 01910.Na and upon activity that has been observed in other clinical trials with ON 01910.Na in patients with MDS.

DETAILED DESCRIPTION:
This is a phase 2, study in which 14 MDS patients with Trisomy 8 or classified as Intermediate-1, -2 and High risk who meet all other inclusion/exclusion criteria will receive ON 01910.Na 800 mg/m^2/24h as an continuous intravenous infusion (CIV) over 48 hours once a week for 3 weeks of a 4-week cycle. As of Amendment 3 to the Protocol, the regimen is changed to 1800 mg/24h for 72 hours every other week for the first four 2-week cycles and every 4 weeks afterwards. The total study duration is 31 weeks, which includes a 2-week screening phase, a 27-week dosing phase, and a 4-week follow-up phase that begins after the last dose of ON 01910.Na. Beginning at week 4, and every 2 weeks thereafter, patients will be assessed for response. Patients who drop out for any reason will not be replaced. Patients who achieve by week 29 a complete or partial response or stabilization of their disease are eligible to receive an additional 24 weeks of ON 01910.Na 1800 mg/24 h over 72 hours per week of a 4-week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS confirmed within 2 weeks prior to study entry according to the World Health Organization (WHO) Criteria or the French-American-British (FAB) Classification.
* Trisomy 8 cytogenetics (simple or combined to other karyotypes) or patient classified as Intermediate-1 with bone marrow blasts equal to or greater than 5%, Intermediate-2 or High Risk MDS according to the IPSS score, or Patients with peripheral blood blasts equal to or greater than 5%.
* At least one cytopenia (Absolute Neutrophil Count < 1800/µl or Platelet Count <100,000/µl or Hemoglobin < 10 g/dL).
* Failure of, or insufficient response to Azacytidine or Decitabine administered for 4 to 6 cycles in patients classified as Intermediate-2 or High risk or to Erythrocyte stimulating agents (failure or insufficient response defined as transfusion dependence or Hemoglobin remaining below 10 g/dl) in Low or Intermediate-1 Risk Trisomy 8 patients.
* Failed to respond to, relapsed following, or opted not to participate in bone marrow transplantation.
* Off all other treatments for MDS (including filgrastim (G-CSF) and erythropoietin) for at least four weeks. As an exception, filgrastim (G-CSF) can be used before, during and after the protocol treatment for patients with documented febrile neutropenia (< 500/µl).
* ECOG Performance Status 0, 1 or 2.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Patient (or his/her legally authorized representative) must have signed an informed consent document indicating that he/she understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

* Anemia due to factors other than MDS (including hemolysis or gastrointestinal bleeding).
* Hypoplastic MDS (cellularity <10%).
* Any active malignancy within the past year except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast.
* History of HIV-1 seropositivity.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Active infection not adequately responding to appropriate therapy.
* Total bilirubin > 1.5 mg/dL not related to hemolysis or Gilbert's disease, ALT or AST > 2 X ULN.
* Serum creatinine > 2.0 mg/dL or calculated creatinine clearance < 60 ml/min/1.73 m^2.
* Ascites requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of <134 Meq/L).
* Women patients who are pregnant or lactating; Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol; Patients who do not agree to use adequate contraceptive [including prescription oral contraceptives (birth control pills), contraceptive injections, intrauterine device (IUD), double-barrier method (spermicidal jelly or foam with condoms or diaphragm), contraceptive patch, or surgical sterilization] before entry and throughout the study; Female patients with reproductive potential who do not have a negative serum beta-HCG pregnancy test at screening.
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.
* Uncontrolled hypertension (defined as a systolic pressure equal to or greater than 160 mmHg and/or a diastolic pressure equal to or greater than 110 mmHg).
* New onset seizures (within 3 months prior to the first dose of ON 01910.Na) or poorly controlled seizures
* Any concurrent investigational agent or chemotherapy, radiotherapy or immunotherapy.
* Treatment with standard MDS therapies or investigational therapy within 4 weeks of starting ON 01910.Na.
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 29 weeks
  The Overall Response Rate is defined as the proportion of patients who achieve a Complete Response, a Partial Response, A Complete Bone Marrow Response or a Hematologic Improvement (HI) according to the 2006 International Working Group (IWG) criteria.
Number of patients with adverse events | From date of signing informed consent until 30 days after last dose of study drug up to 29 weeks
  The NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 will be used to determine the grade of adverse events.

SECONDARY OUTCOMES:
Time to Overall Response | 29 weeks
  Time to Overall Response is calculated from date of first study drug administration to date of first occurrence of any of the following responses: Complete Response (CR), Partial Response (PR), Marrow Complete Response (BMCR) or Hematologic Improvement (HI) as defined by the 2006 International Working Group (IWG) criteria.
Duration of Response | 29 weeks
  Duration of response is calculated from date of first occurrence of any of the following responses: Complete Response (CR), Partial Response (PR), Marrow Complete Response (BMCR) or Hematologic Improvement (HI) as defined by the 2006 International Working Group (IWG) criteria) until the date of disease progression. Patients who did not have disease progression are censored at the last bone marrow or bone marrow morphology assessment date.
Bone Marrow Complete Response | Weeks 5, 13, 21 and 29
  The proportion of patients who achieve a Bone Marrow Complete Response (BMCR) according to 2006 International Working Group (IWG) criteria. Bone marrow blasts are determined in bone marrow differential count.
Cytogenetic Response | 29 weeks
  Cytogenetic Response is defined as the number of patients who achieve a cytogenic response according to 2006 International Working Group criteria. Complete response is defined as the disappearance of the chromosomal abnormality without appearance of new ones. Partial response is defined as at least 50% reduction of the chromosomal abnormality.
Neutrophil Response | 29 weeks
  The number of patients who achieve a Neutrophil Response according to 2006 International Working Group (IWG). Neutrophil Response is defined as at least a 100% increase and an absolute increase greater than 0.5 x 10^9/L. Pretreatment values must be less than 1.0 x 10^9/L.
Platelet Response | 29 weeks
  The number of patients who achieve a Platelet Response according to 2006 International Working Group (IWG). Platelet Response is defined as an absolute of greater than or equal to 30 x 10^9 for patients starting with less than 20 x 10^9/L. increase and an absolute increase greater than 0.5 x 10^9/L. Pretreatment values must be less than 1.0 x 10^9/L.
Erythroid Response | 29 weeks
  The number of patients who achieve an Erythroid Response according to 2006 International Working Group (IWG). Erythroid Response is defined as a Hgb increase equal to or greater than 1.5 g/dL and a relevant reduction of units of red blood cells (RBC) transfusions by an absolute number of at least 4 RBC transfusions/8 weeks compared with the pretreatment transfusion number in the previous 8 wells. Only RBC transfusions given for a Hgb of 9.0 g/dL or lower pretreatment will count in the RBC transfusion response evaluation. Pretreatment values of Hgb must be lower than 11 g/dL.
Time to Disease Progression | 29 weeks
  Time to Disease Progression is calculated from date of first dose of study drug administration to date of disease progression recorded on the hematology response assessment clinical report form.
Time to Acute Myeloid Leukemia (AML) Progression | 29 and 53 weeks
  Time to Acute Myeloid Leukemia (AML) Progression is calculated from date of first study drug administration to date of AML progression recorded on the Off Study Summary clinical report form. Patients who do not have AML disease progression are censored at the last bone marrow or bone marrow morphology assessment date.
Overall Survival | 29 and 53 weeks
  Overall Survival is calculated from date of first study drug administration to date of death. In event of no death prior to study termination or data analysis cutoff, overall survival is censored at the last known date patient was alive
Proportion of patients who achieve a Complete Hematologic Response | Up to 29 weeks
  The proportion of patients who achieve a Complete Remission (CR) Hematologic Response according to 2006 International Working Group (IWG) criteria. Bone marrow blasts are determined in bone marrow differential count.
The proportion of patients who achieve a Partial Remission (CR) | Up to 29 weeks
  The proportion of patients who achieve a Partial Remission (PR) Hematologic Response according to 2006 International Working Group (IWG) criteria. Bone marrow blasts are determined in bone marrow differential count.

CONTACTS AND LOCATIONS:
Overall Officials: Peter L. Greenberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

REFERENCES:
- [Result] Seetharam M, Fan AC, Tran M, Xu L, Renschler JP, Felsher DW, Sridhar K, Wilhelm F, Greenberg PL. Treatment of higher risk myelodysplastic syndrome patients unresponsive to hypomethylating agents with ON 01910.Na. Leuk Res. 2012 Jan;36(1):98-103. doi: 10.1016/j.leukres.2011.08.022. Epub 2011 Sep 14. PMID 21924492
- [Result] Silverman LR, Greenberg P, Raza A, Olnes MJ, Holland JF, Reddy P, Maniar M, Wilhelm F. Clinical activity and safety of the dual pathway inhibitor rigosertib for higher risk myelodysplastic syndromes following DNA methyltransferase inhibitor therapy. Hematol Oncol. 2015 Jun;33(2):57-66. doi: 10.1002/hon.2137. Epub 2014 Apr 29. PMID 24777753
- [Result] Navada SC, Silverman LR. The safety and efficacy of rigosertib in the treatment of myelodysplastic syndromes. Expert Rev Anticancer Ther. 2016 Aug;16(8):805-10. doi: 10.1080/14737140.2016.1209413. Epub 2016 Jul 15. PMID 27400247
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.
- See also: Link for Stanford Cancer Center — http://cancer.stanford.edu/